CLINICAL TRIAL: NCT05056376
Title: Effectiveness and Cost-Effectiveness of Fully-Automated Digital vs. Human Coach-Based Diabetes Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00265873; 1R01DK125780-01 (NIH)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes; Hyperglycemia; Glucose, High Blood; Overweight; Prediabetic State; Impaired Glucose Tolerance; Obesity; Weight Loss; Lifestyle, Healthy; Lifestyle Risk Reduction; Lifestyle, Sedentary
Keywords: Prediabetes; Diabetes Prevention Program; DPP; Obesity; Overweight; Physical Activity; Digital; Artificial Intelligence; Weight
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Overweight; Glucose Intolerance; Obesity; Weight Loss; Risk Reduction Behavior; Sedentary Behavior; Motor Activity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully-Automated Digital Diabetes Prevention Program (Experimental): Participants will receive Sweetch Digital Diabetes Prevention Program consists of a smartphone app and bluetooth-enabled digital body weight scale that syncs with the app.
  Interventions: Behavioral: Digital Diabetes Prevention Program (dDPP)
- Human Coach-Based Diabetes Prevention Program (Active Comparator): Participants will attend a total of 16 weekly sessions during months 1 to 6 and 6 sessions during months 7 to 12. These group sessions may be delivered in-person at the local program or remotely using video conferencing. During these sessions, participants will receive information about lifestyle change behaviors focusing on weight loss, physical activity, and nutrition from a trained lifestyle coach.
  Interventions: Behavioral: Human Coach-based Diabetes Prevention Program (hDPP)

INTERVENTIONS:
Behavioral: Digital Diabetes Prevention Program (dDPP) — The Sweetch app is a hyper-personalized mobile digital coach that provides users with tailored recommendations to promote healthy lifestyle behaviors (150 minutes per week of physical activity, weight reduction, and healthy eating habits) to reduce the risk of type 2 diabetes.
  The Sweetch app uses self-tracking and multiple evidence-based persuasive eCoaching strategies. The Sweetch artificial intelligence algorithm delivers just-in-time support and/or adapt recommendations based on the user's response. For example, push notifications will be sent when the algorithm detects that the user is potentially available and able to act upon the recommendation, based on various parameters including location, previous response, calendar availability, and weather, etc.
  Arms: Fully-Automated Digital Diabetes Prevention Program
Behavioral: Human Coach-based Diabetes Prevention Program (hDPP) — The Human Coach-Based Diabetes Prevention Program will consist of a CDC recognized lifestyle change program. Participants will attend a total of 16 weekly sessions during months 1 to 6 and 6 sessions during months 7 to 12. These group sessions may be delivered in-person at the local program or remotely using video conferencing. During these sessions, participants will receive information about lifestyle change behaviors focusing on weight loss, physical activity, and nutrition from a trained lifestyle coach.
  Arms: Human Coach-Based Diabetes Prevention Program

SUMMARY:
The purpose of this research study is to compare the effectiveness of a fully automated digital diabetes prevention program to standard of care human coach-based diabetes prevention programs for promoting clinically meaningful lifestyle changes to reduce the risk of type 2 diabetes in adults with prediabetes.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all participants giving written informed consent will undergo screening to determine eligibility for study entry. At baseline visit (month 0). Participants who meet the eligibility requirements will be randomly assigned in 1:1 ratio to human coach-based diabetes prevention program or digital diabetes prevention program. An equal number of participants will be randomly assigned to both groups (like flipping a coin).

If participants are randomly assigned to receive the human coach-based diabetes prevention program, the participants will be referred to a local Diabetes Prevention Program close to the participants' area. The Diabetes Prevention Program consists of 16 weekly sessions during months 1 to 6 and 6 sessions during months 7 to 12. These group sessions may be delivered in-person at the local program or remotely using video conferencing. During these sessions, participants will receive information about lifestyle change behaviors focusing on weight loss, physical activity, and nutrition from a trained lifestyle coach.

If participants are randomly assigned to receive the digital Diabetes Prevention Program, the participants will receive the Sweetch Digital Health Kit (Sweetch Health, Ltd.) in the mail within approximately 8-12 days of the participants' first study visit. The Sweetch digital health kit consists of a smartphone app and a digital body weight scale that is connected via Bluetooth to the app. The phone app also consists of brief Centers for Disease Control and Prevention (CDC) lessons on type 2 diabetes prevention, which participants will be encouraged to complete.

There will be a total of 3 study visits (baseline, 6 months, and 12 months), each visit includes fingerstick hemoglobin A1C measurement, weight measurement, and completion of several questionnaires. Height will be measured at the first visit. Throughout the 12-month study, participants will be asked to wear a device on the participants' wrist to measure physical activity for 7 consecutive days following the first visit and once every month thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Laboratory evidence of prediabetes, defined as any of the following lab results, in the past year:

  1. Hemoglobin A1C 5.7% to 6.4%
  2. Fasting glucose 100-125 mg/dL
  3. Plasma glucose of 140-199 mg/dL measured 2 hours after a 75 gm glucose load
* Body mass index (BMI) ≥25 kg/m2 (or≥23 kg/m2 for Asians).
* Proficiency in reading English.
* Smartphone user (Android Operating System (OS) 9.0 or iOS 13.3 or newer).
* Plans to reside in recruitment area for the next 12 months (participant's zip code of residence is within ~45 miles of the study recruitment site.

Exclusion Criteria:

* Medical conditions that prevent adoption of moderate physical activity (per primary care clinician).
* Aortic stenosis.
* Unstable cardiac disease (myocardial infarction, heart failure, or stroke in previous 6 months, currently participating in cardiac rehabilitation).
* Has a pacemaker, implantable cardioverter-defibrillator (ICD), or other implanted electronic device.
* Use of any glucose-lowering medications, weight loss medications, or any systemic glucocorticoids within the previous 3 months.
* Active malignancy of any type or diagnosed with or treated for cancer within the past 2 years. Individuals with basal and squamous cell carcinoma of the skin that has been successfully treated will be allowed to participate.
* Diagnosis of diabetes mellitus.
* Pregnancy or planned pregnancy in the next 12 months.
* Anemia.
* Receiving treatment for iron-deficiency anemia, vitamin B12 deficiency, or folate d efficiency.
* Hemoglobinopathy (HbS or HbC disease).
* Blood transfusion in previous 4 months.
* On dialysis or active organ transplant list.
* Treated with erythropoietin.
* Major psychiatric disorder (schizophrenia) or use of antipsychotic medications within the past 1 year.
* Dementia or Alzheimer's disease.
* Diagnosed with an eating disorder (anorexia nervosa, avoidant/restrictive food intake disorder, binge eating disorder, bulimia nervosa, Pica, rumination disorder, other specified or unspecified feeding or eating disorder)
* Diagnosed or self-reported alcohol or substance abuse.
* Known allergy to steel.
* Participation in another clinical trial related to lifestyle management or diabetes prevention.
* Currently attending or attended a diabetes prevention program in the previous 2 years.
* Unwilling to accept random assignments.
* Had bariatric surgery within the 12 months prior randomization or is planning to undergo bariatric surgery during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestoras Mathioudakis, MD MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Reading Hospital - Tower Health, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Data Coordinating Center (Johns Hopkins University) will prepare a de-identified database that is consistent with HIPAA requirements. The de-identified database will include all study research data and will be stored in a repository at Johns Hopkins University (archive.data.jhu.edu) at a time that will coincide with the online publication of the study primary endpoint paper. The repository will contain documentation designed to facilitate use of the database. The documentation prepared for the repository will include a list and timetable for secondary and exploratory papers planned by the study investigators. Access to the database will be restricted to qualified users. Qualified users will include those investigators who submit valid pre-specified hypotheses and certify that they will not use the data for commercial purposes.
Supporting Information: Study Protocol
Time Frame: The study protocol will be submitted for publication within 1 year of the start of enrollment.

REFERENCES:
- [Derived] Mathioudakis N, Lalani B, Abusamaan MS, Alderfer M, Alver D, Dobs A, Kane B, McGready J, Riekert K, Ringham B, Shehadeh A, Vandi F, Wanigatunga AA, Zade D, Maruthur NM; AI-DPP Study Group. An AI-Powered Lifestyle Intervention vs Human Coaching in the Diabetes Prevention Program: A Randomized Clinical Trial. JAMA. 2025 Dec 16;334(23):2079-2089. doi: 10.1001/jama.2025.19563. PMID 41144242
- [Derived] Abusamaan MS, Ballreich J, Dobs A, Kane B, Maruthur N, McGready J, Riekert K, Wanigatunga AA, Alderfer M, Alver D, Lalani B, Ringham B, Vandi F, Zade D, Mathioudakis NN. Effectiveness of artificial intelligence vs. human coaching in diabetes prevention: a study protocol for a randomized controlled trial. Trials. 2024 May 16;25(1):325. doi: 10.1186/s13063-024-08177-8. PMID 38755706
- See also: Study Website — https://www.nestorasmathioudakislab.com/prediabetesresearchstudy

RESULTS

PARTICIPANT FLOW:
Groups:
- Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP): Participants in the AI-DPP group were referred to Sweetch Health, Ltd, and received a digital health kit from within 8-12 days post-randomization, which included a Bluetooth scale and Sweetch app registration instructions. The app delivered personalized push notifications for weight management, physical activity (PA), and nutrition, informed by both actively collected data (e.g., weight measurements, meal logging) and passively collected data (e.g., geolocation, accelerometry). PA was tracked via smartphone or wearable devices, meals were logged through a food library or photo-based detection, and weight was recorded either automatically through the scale or manually.
  The AI used in the Sweetch intervention consisted of a reinforcement learning algorithm that did not employ large language models. It personalized messaging by continuously learning which prompts, timing, and content elicited greater user engagement. The app also delivered location- and goal-specific nutrition education and included gamification elements and educational resources.
- Human Coach-Based Diabetes Prevention Program (Human-DPP): Participants in the Human-DPP group were referred to one of four 12-month accredited lifestyle change programs: Brancati Center and University of Maryland Medical Center (Baltimore, MD), Pottstown Medical Specialists and Montgomery County DPP (Reading, PA). All four participating DPPs had full plus recognition status from the CDC. Due to COVID-19, all sessions transitioned to synchronous distance learning (i.e., group video conferences).
  Trained lifestyle coaches led sessions based on the CDC's PreventT2 curriculum, covering healthy eating, food tracking, PA, behavior modification, and long-term weight management, with an initial core phase (16 weekly sessions) and a remaining core maintenance phase (bi-weekly to monthly sessions) to complete the 12-month intervention. Of note, our study participants joined DPP cohorts that were comprised of standard enrollees who were not participants in our trial.
Period: Overall Study
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Started | 183 | 185
Completed | 151 | 149
Not Completed | 32 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP) | Total
Number analyzed (Participants) | 183 | 185 | 368
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 60.0 [51.0 to 68.0] | 57.0 [50.0 to 63.0] | 58.0 [50.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 139 | 260
  Male | 62 | 46 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 1 | 1
  Race: Asian | 11 | 16 | 27
  Race: Black or African American | 51 | 49 | 100
  Race: White or Caucasian | 114 | 111 | 225
  Race: More than One Race | 3 | 5 | 8
  Race: Other | 4 | 2 | 6
  Race: Declined to Answer | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 176 | 167 | 343
  Ethnicity: Hispanic or Latino | 5 | 15 | 20
  Ethnicity: Declined to Answer | 1 | 1 | 2
  Ethnicity: Unknown | 1 | 2 | 3
Marital Status [Count of Participants; unit: Participants]
  Married/Partnered | 120 | 121 | 241
  Previously Married | 27 | 26 | 53
  Single/Other | 36 | 38 | 74
Educational Attainment [Count of Participants; unit: Participants]
  High School or Less | 23 | 19 | 42
  Some College/Associate's Degree | 38 | 36 | 74
  Bachelor's Degree | 53 | 55 | 108
  Graduate/Professional Degree | 69 | 74 | 143
  Declined to Answer | 0 | 1 | 1
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: Kg/m^2] | 32.2 [28.2 to 35.9] | 32.5 [29.3 to 37.7] | 32.3 [28.5 to 37.1]
Dyslipidemia [Count of Participants; unit: Participants] — Participants with condition are reported
  Participants | 85 | 86 | 171
Hypertension [Count of Participants; unit: Participants] — Participants with condition are reported
  Participants | 82 | 78 | 160
Back Pain [Count of Participants; unit: Participants] — Participants with condition are reported
  Participants | 52 | 44 | 96
Mood Disorder [Count of Participants; unit: Participants] | 39 | 43 | 82
Osteoarthritis [Count of Participants; unit: Participants] — Participants with condition are reported
  Participants | 39 | 32 | 71
Asthma/COPD [Count of Participants; unit: Participants] | 31 | 28 | 59
BMI Classification [Count of Participants; unit: Participants] — Overweight (BMI 25.0 - 29.9 Kg/m^2); Class I Obesity (BMI 30.0 - 34.9 Kg/m^2); Class II Obesity (BMI 35.0 - 39.9 Kg/m^2); Class III Obesity (BMI >= 40.0 Kg/m^2);
  Participants
    Overweight | 55 | 47 | 102
    Class I Obesity | 70 | 57 | 127
    Class II Obesity | 33 | 47 | 80
    Class III Obesity | 25 | 34 | 59
A1C [Mean (Standard Deviation); unit: %] | 5.8 (0.3) | 5.8 (0.3) | 5.8 (0.3)
Actigraph Measured Moderate-to-Vigorous Physical Activity (MVPA) [Median (Inter-Quartile Range); unit: Minutes per Week] — Actigraph-measured MVPA refers to objectively measured moderate-to-vigorous physical activity using a wrist-worn accelerometer. <150 min/week corresponds to not meeting the recommended PA guidelines for prediabetes.
  Minutes per Week | 237.0 [106.0 to 374.0] | 239.0 [104.0 to 462.0] | 237.0 [105.5 to 418.0]
Actigraphy-measured MVPA <150 min/week [Count of Participants; unit: Participants] — Moderate-to-vigorous PA (MVPA) <150 min/week corresponds to not meeting the recommended PA guidelines for prediabetes.
  Participants | 54 | 65 | 119
Diet Quality [Count of Participants; unit: Participants] — Diet quality at baseline was scored using the Starting the Conversation dietary survey, with lower schools indicating healthier dietary patterns. Scores range from 0 to 16, based on responses to 8 items assessing key dietary patterns.
  Participants
    Healthiest Diet (1-5) | 70 | 73 | 143
    Moderately Healthy Diet (6-10) | 50 | 58 | 108
    Least Healthy Diet (11-16) | 63 | 54 | 117

OUTCOME MEASURES:

1. Primary Outcome: Achievement of CDC's Benchmark for Type 2 Diabetes Risk Reduction as a Binary Outcome (Yes/no)
Description: The primary outcome was the CDC-defined diabetes risk reduction benchmark at 12 months (based on the 2021 standards), defined as at least one of the following:
  1. Weight loss of ≥5%.
  2. Weight loss of ≥4% combined with at least 150 weekly minutes of moderate-to-vigorous PA
  3. An absolute decrease of ≥0.2 points in A1C (measured in %). The A1C endpoint was applicable only to participants with baseline A1C of 5.7% to 6.4%. Maintaining an A1C <6.5% throughout the study was also a criterion for the primary outcome.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 183 | 185
Participants | 58 | 59
Statistical Analysis 1: Comparison: Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) vs Human Coach-Based Diabetes Prevention Program (Human-DPP); The primary analysis was conducted in all randomized participants. Those who did not attend the 12-month study visit were classified as not achieving the primary composite outcome, providing a conservative estimate of intervention effectiveness. The risk difference was estimated using binomial regression; Test type: Non-Inferiority — Noninferiority was defined a priori as the lower bound of the one-sided 95% CI for the risk difference being greater than or equal to -15%; p < 0.05, Regression, Logistic

2. Secondary Outcome: Absolute Weight Change
Description: Absolute weight change (kilograms) from baseline to 12 months
Time Frame: At 12 months
Measure: Median (Inter-Quartile Range); unit: Kg
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 151 | 149
Kg | -1.00 [-3.20 to 1.50] | -1.30 [-4.30 to 1.10]

3. Secondary Outcome: Cost-effectiveness as Assessed by the Markov Model
Description: The investigators will compare the cost-effectiveness of the two interventions based on lifetime horizon by constructing a Markov model with model parameters populated from the trial results as well as other published literature. The model will estimate the incremental cost-effectiveness ratio between the two interventions.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Change in Hemoglobin A1C
Description: Change in HbA1C (percentage points) from baseline to 12 months (among participants with baseline HbA1C of 5.7% - 6.4% who completed the 12-month study visit).
Time Frame: At 12 months
Population: Per-protocol analysis included participants with available 12-month outcome data who did not initiate prohibited medications during the trial. Change in A1C analysis was restricted to participants whose baseline A1C at randomization was between 5.7% and 6.4%.
Measure: Median (Inter-Quartile Range); unit: Percentage of Total Hemoglobin
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 106 | 103
Percentage of Total Hemoglobin | 0.0 [-0.2 to 0.1] | -0.1 [-0.2 to 0.1]

5. Secondary Outcome: Percentage Change in Weight
Description: Percentage change in weight from baseline to 12 months
Time Frame: At 12 months
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 151 | 149
percentage change | -1.03 [-3.73 to 1.46] | -1.43 [-4.03 to 1.14]

6. Secondary Outcome: Mean Weekly Moderate-to-vigorous Physical Activity (MVPA)
Description: Average minutes/week of physical activity assessed using blinded Actigraphy (monthly serial consecutive 7-days wear period). If the participant did not wear their monitor for at least 5 of their 7 assigned days, they were considered noncompliant. In this case, the participant was assigned 0 minutes for physical activity for that week.To obtain the average MVPA minutes per week across the study period, the total MVPA minutes per week from all valid wear periods were summed and divided by the number of available wear periods (maximum of 11 post-baseline visits). Specifically, activity intensity was classified as MVPA if the vector magnitude of accelerometer counts per minute was equal to or greater than 3941 (Montoye's cut point).
Time Frame: At 12 months
Measure: Median (Inter-Quartile Range); unit: Minutes per Week
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 151 | 149
Minutes per Week | 210.5 [134.5 to 344] | 174.4 [73.9 to 321.3]

7. Secondary Outcome: Incidence of Diabetes-range A1C
Description: Number of individuals who had an AIC in the diabetes range (A1C ≥6.5%) at the 6-month or 12-month timepoint.
Time Frame: At either 6 or 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 151 | 149
Participants | 8 | 7

8. Secondary Outcome: Acceptability as Assessed by the 32-item Acceptability Questionnaire
Description: To compare the acceptability of the two interventions (satisfaction, utility, interest, motivation, user experience, etc.) using the 32-item acceptability questionnaire.
  Scoring: Sum up all responses to questions 1-31, divide by 155 and multiply by 100 to calculate percentage score out of 100%. The range of possible scores is 20% (lowest acceptability) to 100% (highest possible acceptability).
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

9. Secondary Outcome: Correlation Between Self-reported and Measured Physical Activity
Description: To evaluate the correlation between self-reported PA data collected using different methods:
  * Data collected and reported by hDPPs
  * Self-reported PA data collected by study team obtained at 1-month intervals
  * Objectively measured PA data (Actigraphy) obtained at 1-month intervals
Time Frame: 6 months and 12 months
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: Program Initiation Rate
Description: Program initiators were defined as participants who attended at least one in-person session (Human-DPP) or registered and used the Sweetch app (AI-DPP).
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 183 | 185
Participants | 171 | 153

11. Secondary Outcome: Program Completion Rate
Description: Program completers attended ≥8 sessions in months 1-6 and spanned ≥9 months (Human-DPP), or engaged with the app for ≥8 weeks during months 1-6 with a span of ≥9 months between initiation and last engagement (AI-DPP).
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
Number analyzed (Participants) | 183 | 185
Participants | 117 | 93

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up (12-month visit)
Description: Grade 1: mild, asymptomatic, or mild symptoms; clinical or diagnostic observations only; no intervention required;Grade 2: moderate, requiring minimal or local intervention;Grade 3: severe or medically significant but not immediately life-threatening, necessitating hospitalization or prolongation of hospitalization; disabling; limits self-care activities of daily living;Grade 4: life-threatening consequences requiring urgent intervention;Grade 5: death related to the adverse event.
Arm/Group | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) | Human Coach-Based Diabetes Prevention Program (Human-DPP)
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/185
Serious Adverse Events (participants affected / at risk) | 36/183 | 6/185
Other Adverse Events (participants affected / at risk) | 10/183 | 3/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) (N=183) | Human Coach-Based Diabetes Prevention Program (Human-DPP) (N=185)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3, not related
Fracture of ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 3, not related
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 4, not related
Breast malignant tumors (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) — Grade 3, not related
Phacoemulsification (Eye disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 3 (3) | 0 (0) — Grade 3, not related
Diabetes mellitus (Endocrine disorders) | 1 (1) | 0 (0)
Otalgia (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Grade 3, not related
Flank pain (Renal and urinary disorders) | 2 (3) | 0 (0) — Grade 3, not related
Foot drop (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3, not related
Foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Grade 3, not related
Hammer toe surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Grade 3, not related
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3, not related
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3, not related
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 3, not related
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 3, not related
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 3, not related
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 3, not related
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Grade 3, not related
Meniscus injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 3, not related
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) — Grade 3, not related
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3, not related
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3, not related
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1) — Grade 4, not related
Prostate cancer stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Grade 3, not related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 4, not related
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3, not related
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) — Grade 3, not related
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 3, not related
Stem cell transplant (Surgical and medical procedures) | 1 (1) | 0 (0) — Grade 3, not related
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Grade 3, not related
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3, not related
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) — Grade 3, not related
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3, not related
Wrist operation NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 3, not related
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Intelligence-Based Diabetes Prevention Program (AI-DPP) (N=183) | Human Coach-Based Diabetes Prevention Program (Human-DPP) (N=185)
Anxiety (Psychiatric disorders) | 0 | 1
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalized anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study has limitations. It was unmasked, relied on surrogate outcomes, and DPP delivery may have varied by site. App updates and study visits outside standard DPP exposures may have influenced outcomes. Referrals were not from primary care, and missing data or assumptions about physical activity had minimal sensitivity impacts. COVID-19 altered DPP delivery, and results may not generalize to broader prediabetes populations due to the sample's high activity levels and education.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT05056376/Prot_SAP_000.pdf